CLINICAL TRIAL: NCT00471133
Title: A Phase Ia/Ib Study of the Safety and Immunogenicity of a Xenogeneic Tyrosinase DNA Vaccine Melanoma
Brief Title: Safety and Immunogenicity of a Melanoma DNA Vaccine Delivered by Electroporation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ichor Medical Systems Incorporated (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Drew Hannaman, Ichor Medical Systems, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-003; NCT00466427 (obsolete NCT alias)
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Melanoma (Skin); Intraocular Melanoma
Keywords: melanoma; DNA vaccine; tyrosinase; electroporation
MeSH Terms: conditions — Melanoma; Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xenogeneic Tyrosinase (Experimental)
  Interventions: Biological: Xenogeneic Tyrosinase DNA Vaccine; Device: TriGrid Delivery System for Intramuscular Electroporation

INTERVENTIONS:
Biological: Xenogeneic Tyrosinase DNA Vaccine
Device: TriGrid Delivery System for Intramuscular Electroporation

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a DNA vaccine encoding a melanosomal antigen in melanoma patients at risk for disease progression or recurrence. In this study, the vaccine will be administered intramuscularly using a device that applies brief electrical fields to the tissue at the site of injection (a technique known as electroporation). It is expected that this device will improve the delivery of the vaccine. This study is being performed to determine if this procedure can be administered safely and if it is capable of inducing immune responses to the vaccine.

DETAILED DESCRIPTION:
This study is designed to evaluate administration of a xenogeneic DNA vaccine encoding the melanosomal antigen tyrosinase by in vivo electroporation in patients with malignant melanoma. The objectives of the study are to characterize the safety and immunogenicity of a DNA vaccine encoding the murine tyrosinase gene delivered administered intramuscularly using the electroporation based TriGrid Delivery System (Ichor Medical Systems). We will assess the nature, frequency, and severity of any toxicity associated with vaccination at escalating pINGmuTyr doses and then expand enrollment at then expand enrollment at the Maximum Tolerated Dose to assess immunologic responses to the tyrosinase antigen.

The hypotheses being tested are that the procedure is feasible and safe and that it induces immune responses specific for tyrosinase in patients with stage IIB-IV malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented, histologically confirmed malignant melanoma, American Joint Commission on Cancer (AJCC) Stage IIB- IV. Patients with stage IIb-III disease are only eligible after standard surgical care with wide local excision and appropriate lymph node sampling. Patients with stage IIb, IIc, or III melanoma who are free of disease after surgical resection are also eligible, only if they have refused high dose Interferon-alfa (INTRON A) or have had a recurrence while on Interferon-alfa.
* Patients with choroidal melanoma may participate if they fulfill one of the following criteria: Basal diameter >16mm; Height >8mm or involvement of the ciliary body with tumor.
* Patients must be at least 18 years of age and must be capable of understanding the consent form and giving informed consent.
* Karnofsky Score > 80
* Life Expectancy > 6 months
* HLA-A1, A2, A24, or B35+ as assessed by low resolution phenotyping
* White blood cell count ≥ 2,000/mm3
* Platelet count ≥ 100,000/mm3
* Neutrophil count ≥ 1,000/mm3
* Hemoglobin ≥ 9.0 g/dL
* Serum AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Serum Bilirubin ≤ 2.0 mg/dL
* Serum Creatinine ≤ 2.0 mg/dL
* Serum Alkaline Phosphatase < 2.5 times ULN
* Serum Creatine phosphokinase (CPK) < 2.5 times ULN

Exclusion Criteria:

* Documented metastases in brain
* Clinical history of HIV, HepB, HepC, and/or HTLV I.
* Active autoimmune disease other than vitiligo
* Patients previously immunized using the tyrosinase DNA sequence, protein, or peptides.
* Systemic immunosuppressive therapy (corticosteroids, or other immunosuppressive drugs) within the previous 28 days
* Surgery and/or radiotherapy within the previous 28 days
* Chemotherapy and/or biotherapy within the previous 28 days
* Participation in an investigational study within previous 28 days
* Patients with cardiac demand pacemakers.
* Women who are pregnant or < 3 months post partum or nursing.
* Women of child-bearing potential and sexually active men must be using appropriate contraception during the course of this study.
* Any other concurrent medical condition that in the opinion of the Principal Investigator or co-Principal Investigator's would preclude study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and feasibility of electroporation mediated intramuscular delivery of a mouse tyrosinase plasmid DNA vaccine in patients with stage IIB, IIC, III, or IV melanoma. | one year

SECONDARY OUTCOMES:
Assess patients with measurable tumor for evidence of anti-tumor response following immunization. | 6 months
Assess the magnitude and frequency of tyrosinase specific immunologic responses in the immunized patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jedd D. Wolchok, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Yuan J, Ku GY, Adamow M, Mu Z, Tandon S, Hannaman D, Chapman P, Schwartz G, Carvajal R, Panageas KS, Houghton AN, Wolchok JD. Immunologic responses to xenogeneic tyrosinase DNA vaccine administered by electroporation in patients with malignant melanoma. J Immunother Cancer. 2013 Nov 18;1:20. doi: 10.1186/2051-1426-1-20. eCollection 2013. PMID 24829756